CLINICAL TRIAL: NCT06942156
Title: A Prospective, Multicenter, Open-Label, Randomized, Comparative, Phase 4 Trial to Optimize Immunosuppressive Therapy Using Everolimus and Low-dose Calcineurin Inhibitors in Heart Transplant Patients in Korea
Brief Title: Optimize Immunosuppressive Therapy Using Everolimus and Low-dose Calcineurin Inhibitors in Heart Transplant Patients in Korea
Acronym: OPTIMIZE-HTx
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B95_05HTx2501
Record Dates: First submitted 2025-04-11; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Heart Transplant
Keywords: Heart transplant; Everolimus
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Certirobell Tablet (Experimental): Everolimus
  Interventions: Drug: Everolimus
- Myrept Tablet/Capsule (Active Comparator): Mycophenolate mofetil
  Interventions: Drug: Mycophenolate mofetil Tablet/Capsule

INTERVENTIONS:
Drug: Everolimus — Up to 1.5g BID(total 3g daily), PO - Check the blood concentration of Everolimus at each visit
  Other Names: Certirobell Tablet
  Arms: Certirobell Tablet
Drug: Mycophenolate mofetil Tablet/Capsule — Up to 1.5g BID(total 3g daily), PO
  Other Names: Myrept® Cap./Tab.
  Arms: Myrept Tablet/Capsule

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lower dose calcineurin inhibitors (CNI) in combination with Everolimus in Korean heart transplant recipients.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, randomized, comparative, phase 4 trial to optimize immunosuppressive therapy using everolimus and low-dose calcineurin inhibitors in heart transplant patients in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Patients with stable heart transplant graft function at least 28~100 days post transplant.
3. Patients who are appropriate for combination therapy with Everolimus and Calcineurin inhibitor (CNI) at the investigator's discretion

Exclusion Criteria:

1. Recipients who have had a prior organ transplant, or who underwent a heart transplant with the simultaneous transplantation of another organ.
2. Recipients of heart from ABO-incompatible donor
3. Recipients of heart from the donor aged 70 or older

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-14 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
hierarchical composite assessed using the win-ratio | baseline, 12 months
  hierarchical composite assessed using the win-ratio, including graft survival, treated rejection episodes, change in percent atheroma volume, and change in eGFR.

SECONDARY OUTCOMES:
Graft rejection | Baseline and 6, 12 months after drug administrations
  Time to onset of Graft rejection
Newly developed Graft dysfunction | Baseline and 6, 12 months after drug administrations
  Frequency of incidence
Change in renal function | Baseline and 6, 12 months after drug administrations
  Change in eGFR
CAV ISHLT grade | Until 12 months
  Coronary Arterial Vasculopathy(CAV) assessed by ISHLT grade for CAV (ISHLT: International Society for Heart and Lung Transplantation)
  * CAV0 (Not significant): No detectable angiographic lesion
  * CAV1 (Mild): Angiographic LM<50% or Primary vessel with maximum lesion<70% or Branch stenosis<70%
  * CAV2 (Moderate): Angiographic LM<50%, Single primary vessel≥70% or Isolated branch stenosis in 2 system≥70%
  * CAV3 (Severe): Angiographic LM≥50% or ≥2 primary vessels ≥70% or Isolated branch stenosis in all 3 system≥70% or CAV1 or CAV2 with allograft dysfunction (LVEF≤45%) or evidence of significant restrictive physiology

CONTACTS AND LOCATIONS:
Overall Officials: Jin-O Choi, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No